CLINICAL TRIAL: NCT05429138
Title: Ovarian Reserve and Semen Parameters Evolution During Adjuvant Therapy in Melanoma
Acronym: MELpreserv
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-A02601-40
Record Dates: First submitted 2022-05-12; First posted 2022-06-23 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Melanoma
Keywords: melanoma; ovarian reserv; semen parameters; fertility; adjuvant
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and semen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Immunotherapy cohort: Patient that received adjuvant immunotherapy
  Interventions: Other: biological sampling
- Targeted therapy: Patient that received adjuvant targeted therapy
  Interventions: Other: biological sampling

INTERVENTIONS:
Other: biological sampling — Biological sampling: blood and semen

SUMMARY:
Prospective multicentric study including women aged 18 to 37 and men aged 18 to 45 during their visit to centers for the study and storage of human sperm and eggs (CECOS). Subjects will be included before adjuvant treatment initiation (T0) and immediately after treatment (approximately 1 year after initiation, T1), and, in late post treatment (1 year after treatment cessation, T2).

Expected results: This study will evaluate the evolution of AMH, AFC, and semen parameters in our cohort of melanoma patients treated with anti-PD-1 and targeted therapy in an adjuvant and neoadjuvantsettings.

DETAILED DESCRIPTION:
To the best of our knowledge, no data is available in humans on the impact of anti-PD-1 immunotherapies and therapies targeting the MAP kinase pathway, in adjuvant settings, on ovarian reserve and semen quality.

Main objective: to measure pre-treatment (T0) and immediate post-treatment (T1) evolution of anti-Müllerian hormone (AMH) levels reflecting the ovarian reserve in women, and of the total motile sperm count per ejaculate in men, in patients of childbearing age treated with anti-PD-1 immunotherapy or targeted therapies in an adjuvant situation for melanoma at high risk of recurrence.

Method: Prospective multicentric study including women aged 18 to 37 and men aged 18 to 45 during their visit to centers for the study and storage of human sperm and eggs (CECOS). Subjects will be included before adjuvant treatment initiation (T0) and immediately after treatment (approximately 1 year after initiation, T1), and, in late post treatment (1 year after treatment cessation, T2).

At each of their visit to CECOS (T0, T1 and T2), the women will have an AMH assay and an antral follicle count (AFC) by ultrasound while the men will perform a semen analysis (count, spermocytogram and staining with aniline blue for analysis of chromatin condensation).

A standardized questionnaire aimed at collecting data about factors that may alter fertility will be submitted at each of these visits.

Expected results: This study will evaluate the evolution of AMH, AFC, and semen parameters in our cohort of melanoma patients treated with anti-PD-1 and targeted therapy in an adjuvant settings.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have provided a signed, dated and written consent prior to any specific procedures, sampling and analyses
* Patients with valide Health Inssurance Scheme
* Female between 18 and 37 years old and male between 18 and 45 years old
* During the 2 months before the introduction of an approved regimen of adjuvant anti-PD-1 immunotherapy or neoadjuvant plus adjuvant or targeted therapy for an high-risk of reccurence melanoma
* Adjuvant or neoadjuvant plus adjuvant treatment must be prescribed as part of routine care

Exclusion Criteria:

* Individuals deprived of liberty or placed under the authority of a tutor
* Patients unable to understand, read and/or sign an informed consent
* History of cytotoxic treatment before T0 that can alterate the studied parameters
* In male, totale motile sperm count per ejaculate inferior to 39 millions at T0
* In women, an age-specific AMH level inferior to the 10th percentile at T0
* Any condition which in the Investigator's opinion would jeopardize compliance with the protocol of the study
* Patients that will received an investigational treatment during the study timeframe (an observational research is allowed)
* Patients who have changed the type of adjuvant treatment during adjuvant treatment (targeted switch therapy versus targeted immunotherapy and vice versa) or after the neoadjuvant phase due to the pathological response obtained.

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: Patients of childbearing age treated with an adjuvant anti-PD-1 immunotherapy or neoadjuvant plus adjuvant or targeted therapies for a melanoma at high risk of recurrence
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-12-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
measurement of biological parameters : Anti-Müllerian hormone (AMH) levels in women | T1 (=Day0 + 12 months)
  change in Anti-Müllerian hormone (AMH) levels in women
measurement of biological parameters : Change in sperm motility count in men | T1 (=Day0 + 12 months)
  Change in sperm motility count per ejaculate in men

SECONDARY OUTCOMES:
measurement of biological parameters : Antral follicle count in women | T0 = Day 0 = treatment initiation; T1 = Day0 + 12 months; T2 = T1 + 12 months.
  change in antral follicle count in women
measurement of biological parameters : levels of spermatozoids with sperm chromatin abnormalities | T0 = Day 0 = treatment initiation; T1 = Day0 + 12 months; T2 = T1 + 12 months.
  change of rate of spermatozoids with sperm chromatin abnormalities
measurement of biological parameters : Change in sperm count | T0 = Day 0 = treatment initiation; T1 = Day0 + 12 months; T2 = T1 + 12 months.
  Change in sperm count (spermogram) during time
measurement of biological parameters : Change in sperm motility count | T0 = Day 0 = treatment initiation; T1 = Day0 + 12 months; T2 = T1 + 12 months.
  Change in sperm motility count (spermogram)

OTHER OUTCOMES:
measurement of biological parameters : change in sperm morphology | T0 = Day 0 = treatment initiation; T1 = Day0 + 12 months; T2 = T1 + 12 months.
  change in sperm morphology (using spermogram)

CONTACTS AND LOCATIONS:
Overall Officials: Nausicaa Malissen, MD, PhD, Principal Investigator — AP-HM
Locations (12):
- France (12):
  - CHU de Bordeaux, Bordeaux
  - AP-HM, Marseille
  - Hôpital Saint-Joseph, Marseille
  - CHU Montpellier, Montpellier
  - CHU de Nantes, Nantes
  - CHU NICE L'archet, Nice
  - CHRU de Nîmes, Nîmes
  - APHP- Ambroise Paré, Paris
  - APHP-Cochin, Paris
  - APHP-Saint Louis, Paris
  - Oncôpole de Toulouse, Toulouse
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No